CLINICAL TRIAL: NCT00357110
Title: A Randomised Phase II Study Comparing Anastrozole and Fulvestrant to Anastrozole for Adjuvant Treatment of Postmenopausal Patients With Early Breast Cancer and Disseminated Tumour Cells in Bone Marrow
Brief Title: Anastrozole and Fulvestrant Compared to Anastrozole as Adjuvant Treatment of Postmenopausal Patients With Breast Cancer
Acronym: @FAME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6990C00001; ABCSG21; Eudract No 2005-005715-22
Record Dates: First submitted 2006-07-20; First posted 2006-07-27 (Estimated); Results first posted 2010-01-22 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Breast Cancer
Keywords: Breast neoplasms; breast cancer; early breast cancer; oncology; cancer; breast cancer micrometastasis; fulvestrant
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Fulvestrant; Anastrozole

ARMS (2):
- 1 (Active Comparator): Anastrozole monotherapy
  Interventions: Drug: Anastrozole
- 2 (Experimental): Anastrozole + Fulvestrant
  Interventions: Drug: Fulvestrant; Drug: Anastrozole

INTERVENTIONS:
Drug: Fulvestrant — intramuscular injection
  Other Names: Faslodex; ZD9238
  Arms: 2
Drug: Anastrozole — 1 mg oral tablet
  Other Names: Arimidex; ZD1033

SUMMARY:
Purpose is to compare the frequency of events (presence of Disseminated Tumour Cells, clinical recurrence and/or death) after 1 and 2 years of adjuvant treatment with anastrozole and fulvestrant or anastrozole alone in patients with early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with hormone receptor-positive early breast cancer and a positive Disseminated Tumour Cell immunocytochemical result from bone marrow aspiration prior to randomisation

Exclusion Criteria:

* Inflammatory and/or metastatic breast cancer.
* Current or previous malignancy within previous 5 years (other than Breast cancer or adequately treated non-melanoma skin cancer or in-situ cervical cancer).
* History of bleeding diathesis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Breast Cancer Established Brands Team Medical Science Director, MD, Study Director — AstraZeneca
Locations (25):
- Austria (10):
  - Research Site, Feldkirch
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Leoben
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Sankt Veit im Pongau
  - Research Site, Vienna
  - Research Site, Wiener Neustadt
- Germany (7):
  - Research Site, Bayreuth
  - Research Site, Essen
  - Research Site, Hamburg-Eppendorf
  - Research Site, Heidelberg
  - Research Site, Munich
  - Research Site, Rostock
  - Research Site, Tübingen
- Norway (8):
  - Research Site, Drammen
  - Research Site, Fredrikstad
  - Research Site, Kristiansand
  - Research Site, Oslo
  - Research SIte, Porsgrunn
  - Research Site, Stavanger
  - Research Site, Trondheim
  - Research Site, Tønsberg

RESULTS

PARTICIPANT FLOW:
Groups:
- Fulvestrant + Anastrozole: fulvestrant 500 mg + anastrozole 1 mg
- Anastrozole: anastrozole 1 mg
Period: Overall Study
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Started | 6 | 7
Completed | 1 | 2
Not Completed | 5 | 5
Not completed — Early study termination | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant + Anastrozole | Anastrozole | Total
Number analyzed (Participants) | 6 | 7 | 13
Age Continuous [Mean (Standard Deviation); unit: age in years at baseline] | 60.5 (5.4) | 63.4 (3.5) | 62.1 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patients Event-free at 12 Months (Where Event = Death (From Any Cause), Disseminated Tumour Cells (DTC) Positive at 12 Months or Clinical Disease Recurrence)
Description: Number of patients event-free
Time Frame: 12 month period following randomisation
Measure: Number; unit: Participants
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 6 | 7
Participants | 6 | 7

ADVERSE EVENTS:
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/7
Other Adverse Events (participants affected / at risk) | 5/6 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant + Anastrozole (N=6) | Anastrozole (N=7)
Goitre (Endocrine disorders) | 0 | 1
Haemorrhoid Operation (Gastrointestinal disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Varicose Vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant + Anastrozole (N=6) | Anastrozole (N=7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 2 | 1
Hot Flush (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Unevaluable Event (General disorders) | 2 | 1
Fatigue (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Injection Site Pruritus (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 0
Depressed Mood (Psychiatric disorders) | 1 | 0
Mood Altered (Psychiatric disorders) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Weight Decreased (Investigations) | 1 | 0
Weight Increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Renal Pain (Renal and urinary disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Keratitis Herpetic (Infections and infestations) | 1 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will provide ASTRAZENECA as soon as possible with preliminary data and drafts of proposed results communications and with the proposed final draft at least 14 days prior to submission of an abstract and 30 days prior to submission of a manuscript. ASTRAZENECA can, upon written request, embargo communications regarding trial results for no more than 45 days from the date of the written request. ASTRAZENECA cannot require changes to the communication and cannot extend the embargo.